CLINICAL TRIAL: NCT05244798
Title: Neoadjuvant Chemotherapy or Neoadjuvant Chemoradiotherapy Plus Sintilimab Versus Neoadjuvant Chemoradiotherapy for Locally Advanced Esophageal Squamous Cell Carcinoma: a Multicenter, Randomized, Controlled, Phase III Trial
Brief Title: Sintilimab Plus NCT or NCRT Versus NCRT for ESCC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Hebei Medical University Fourth Hospital (Other); Anhui Provincial Hospital (Other Government); The First Affiliated Hospital with Nanjing Medical University (Other); Anyang Tumor Hospital (Other); Shantou Central Hospital (Other); Innovent Biologics (Suzhou) Co. Ltd. (Industry); GeneCast Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yongtao Han, Chief of Thoracic Surgery, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCCH-TS2201
Record Dates: First submitted 2022-01-30; First posted 2022-02-17 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — sintilimab; Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group of sintilimab combined with neoadjuvant chemotherapy (Experimental): sintilimab (D1 administration) was given in combination with chemotherapy (TP regimen: albumin-paclitaxel + carboplatin, D1 administration) for 2 cycles. Every 3 weeks, there was a dosing cycle (Q3W). Surgery was performed 6-8 weeks after completion of neoadjuvant therapy. If the patients without vital tumor cells in primary and lymph nodes after surgery, they only need regular follow-up visit. If the patients with non-pCR resected, those patients need to receive adjuvant immunotherapy. And if the patients with non-R0 resected, the regimen of those patients need to carefully decide based on multidisciplinary team discussed.
  Interventions: Drug: Sintilimab; Drug: Chemotherapy
- Group of sintilimab combined with neoadjuvant chemoradiotherapy (Experimental): sintilimab (D1) was administered in combination with concurrent chemoradiotherapy. Chemotherapy regimen: TP regimen: albumin-paclitaxel + carboplatin, D1 administration, 2 cycles. Every 3 weeks, there was a dosing cycle (Q3W). Radiotherapy regimen: according to IMRT treatment plan, the total dose was 41.4Gy, divided into 23 times, 5 days a week. Surgery was performed 6-8 weeks after completion of neoadjuvant therapy. If the patients without vital tumor cells in primary and lymph nodes after surgery, they only need regular follow-up visit. If the patients with non-pCR resected, those patients need to receive adjuvant immunotherapy. And if the patients with non-R0 resected, the regimen of those patients need to carefully decide based on multidisciplinary team discussed.
  Interventions: Drug: Sintilimab; Radiation: radiotherapy; Drug: Chemotherapy
- Group of neoadjuvant chemoradiotherapy (Other): The control group received neoadjuvant chemoradiotherapy and the regimen was as follows:Chemotherapy regimen: TP regimen: albumin paclitaxel + carboplatin, D1 administration, 2 cycles. Every 3 weeks, there was a dosing cycle (Q3W). Radiotherapy regimen: according to IMRT treatment plan, the total dose was 41.4Gy, divided into 23 times, 5 days a week. Surgery was performed 6-8 weeks after completion of neoadjuvant therapy. If the patients without vital tumor cells in primary and lymph nodes after surgery, they only need regular follow-up visit. If the patients with non-pCR resected, those patients need to receive adjuvant immunotherapy. And if the patients with non-R0 resected, the regimen of those patients need to carefully decide based on multidisciplinary team discussed.
  Interventions: Radiation: radiotherapy; Drug: Chemotherapy

INTERVENTIONS:
Drug: Sintilimab — Sintilimab: D1 administration) for 2 cycles. Every 3 weeks was a dosing cycle (Q3W)
  Arms: Group of sintilimab combined with neoadjuvant chemoradiotherapy; Group of sintilimab combined with neoadjuvant chemotherapy
Radiation: radiotherapy — Radiotherapy: According to IMRT treatment plan, the total dose was 41.4Gy, divided into 23 times, 5 days a week.
  Arms: Group of neoadjuvant chemoradiotherapy; Group of sintilimab combined with neoadjuvant chemoradiotherapy
Drug: Chemotherapy — Neoadjuvant chemotherapy with TP regimen: albumin-paclitaxel + carboplatin, D1 administration) for 2 cycles. Every 3 weeks was a dosing cycle (Q3W).

SUMMARY:
Comparative analysis of patients with resectable locally advanced esophageal squamous cell carcinoma treated with neoadjuvant chemotherapy or neoadjuvant chemoradiotherapy combined sintilimab versus neoadjuvant chemoradiotherapy.

DETAILED DESCRIPTION:
The research process is divided into three stages: firstly, the stage of screening period for 14 days. Qualified subjects will enter the treatment period after completion of screening examination and evaluation. And then, the stage of treatment period: Experimental group (group A) received sintilimab combined with neoadjuvant chemotherapy regimen: preoperative neoadjuvant, sintilimab (D1 administration) combined with chemotherapy (TP regimen: albumin-paclitaxel + carboplatin, D1 administration) for 2 cycles. Every 3 weeks, there was a dosing cycle (Q3W). The experimental group (group B) received neoadjuvant sintilimab combined concurrent chemoradiotherapy: preoperative sintilimab (D1 administration) combined with neoadjuvant concurrent chemoradiotherapy. Chemotherapy regimen: TP regimen: albumin-paclitaxel + carboplatin, D1 administration, 2 cycles. Every 3 weeks, there was a dosing cycle (Q3W). Radiotherapy regimen: according to IMRT treatment plan, the total dose was 41.4Gy, divided into 23 times, 5 days a week. And the control group (group C) received neoadjuvant chemoradiotherapy and the regimen was similar with group B. Surgery was performed 6-8 weeks after completion of neoadjuvant therapy. If the patient without vital tumor cells in primary and lymph nodes after surgery, they only need regular follow-up visit. If the patients with non-pCR resected, those patients need to receive adjuvant immunotherapy. And if the patients with non-R0 resected, the regimen of those patients need to carefully decide based on multidisciplinary team discussed. Lastly, the stage of postoperative assistance, the researchers selected postoperative treatment according to the guidelines for the diagnosis and treatment of esophageal cancer. Patients were followed up for efficacy and safety within 90 days after surgery, once every 3 months for 2 years and once every 6 months for 2-5 years.

ELIGIBILITY:
Inclusion criteria:

1. Aged 18 to 75, both sexes;
2. Patients with histologically confirmed locally advanced (cT1N2-3M0 or cT2-4aN0-3M0) thoracic esophageal squamous cell carcinoma (8th UICC-TNM stage);
3. Cervical contrast-enhanced CT showed no suspicious metastatic lymph nodes. Imaging examination showed no systemic metastasis.
4. R0 resection is expected to be achieved;
5. Physical state ECOG 0 ~ 1;
6. No previous antitumor therapy for esophageal cancer, including chemotherapy, radiotherapy (including radiotherapy planned during the study), hormone therapy, and immunotherapy;
7. Measurable lesions (according to RECIST v1.1);
8. There was no operation contraindications in the evaluation of various organ functions before operation;
9. The following laboratory tests confirm that the bone marrow, liver and kidney functions meet the requirements for study participation:

   * Hemoglobin ≥90g/L;
   * White blood cell count ≥ lower limit of laboratory normal;
   * Neutrophil absolute value (ANC) ≥1.5×109/L;
   * Platelet count ≥100×109/L; Total bilirubin ≤1.5× upper limit of normal (ULN);
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN;
   * Prothrombin time ≤16 seconds and international normalized ratio ≤1.5×ULN; Creatinine ≤1.5×ULN or Cr clearance ≥50 mL/min (calculated using Cockcroft-Gault formula);
10. Fertile women must consent to use effective contraception (e.g. intrauterine devices, birth control pills, or condoms) during the study medication period and within 60 days of the last study medication, have a negative serum pregnancy test within 7 days before study enrollment, and be non-lactating; Men agree that they must use effective contraception during the study medication period and for 60 days after the last study medication;
11. The informed consent must be understood and signed.

Exclusion criteria:

Patients who met any of the following criteria were excluded from the study:

1. Malignant tumors other than esophageal cancer (cured localized tumors, including cervical carcinoma in situ, skin basal cell carcinoma and prostate carcinoma in situ, were not excluded) had occurred within 5 years before randomization; Prostate cancer patients receiving hormone therapy with DFS for more than 5 years were not excluded).
2. Patients with high blood tendency who had a history of gastrointestinal bleeding within 6 months before randomization, or had coagulopathy at the time of enrollment, or were receiving thrombolysis or anticoagulant therapy;
3. Severe cardiovascular and cerebrovascular diseases:

   • New York Heart Association (NYHA) class II or higher congestive heart failure, unstable angina, myocardial infarction, poorly controlled arrhythmias, or cerebrovascular accidents within 12 months before randomization.

   LVEF (left ventricular ejection fraction) <50% on echocardiography. Corrected QT interval (QTc) >480ms (calculated using Fridericia's method; if QTc was abnormal, three consecutive tests were performed at 2 min intervals and the mean value was taken).

   Medically difficult to control hypertension (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100mmHg) (based on the average of ≥2 measurements).

   • A previous hypertensive crisis or hypertensive encephalopathy.
4. Previous history of interstitial lung disease or pneumonia requiring steroid treatment at enrollment;
5. Had active tuberculosis at the time of randomization, or had received anti-tuberculosis therapy within 1 year before randomization;
6. Asthma at random requiring intermittent use of bronchodilators or other medical interventions;
7. Patients with infectious diseases requiring systemic treatment (oral or intravenous administration) within 4 weeks before randomization; for active hepatitis, effective treatment was required before enrollment;
8. Severe unhealed wounds, active ulcers, and untreated fractures at random;
9. Combined with other inoperable conditions;
10. The previous operation resulted in the inability to use stomach instead of esophagus to reconstruct the digestive tract in this operation;
11. Was receiving systemic steroid therapy (more than 10mg of prednisone daily or equivalent) or other immunosuppressive agents during the 2 weeks prior to randomization;
12. Severe allergy to chemotherapy drugs (albumin paclitaxel or cisplatin) or any monoclonal antibody;
13. Has had an active autoimmune disease requiring systemic treatment (i.e., immunomodulatory drugs, corticosteroids, or immunomodulatory drugs) in the past 2 years; However, replacement therapy (e.g., thyroxine, insulin, or replacement therapy with physiologic corticosteroids for adrenal or pituitary insufficiency) is not considered systemic therapy and is allowed for use and enrollment;
14. Previous organ transplant recipients;
15. If HBsAg(+) and/or HBcAb(+) are required, HBV DNA must be < 500IU/mL. (If the lower limit of the local center's minimum detectable value is higher than 500IU/mL, after discussion with the sponsor, Enrollment was determined on a case-to-case basis) and continued to receive effective anti-HBV therapy that was already in use during the study period, or entecavir or tenofovir therapy was started prior to study medication;
16. Hcv-rna testing should be performed if HCV antibody is positive, and HCV-RNA>10^3 copy number /mL should be excluded;
17. Co-infection with HIV;
18. In the judgment of the investigator, there are other circumstances that are not suitable for participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathology complete response rate, pCR | 3 months after the surgery
  Definition of pathology complete response is "no cancer cell, including lympho nodes" which corresponds with tumor regression score 0 definition of pathologic response is as follows. Tumor regression score Grade 0 and 1 will be defined as "responder" and 2 and 3 will be considered as "non-responders".

SECONDARY OUTCOMES:
Treatment related adverse event, TRAE | 3 months after the surgery
  The TRAE defined as the proportion of participants who have treatment-related adverse events assessed by National Cancer Institute Common Terminology Criteria for Adverse Event, Version 4.0 (CTCAE v4.0).
Major Pathological Remission rate, MPR | 3 months after the surgery
  The residual tumor after neoadjuvant treatment ≤ 10% residual tumor lesion in surgical specimen compared to baseline.
Rate of R0 resection | 3 months after the surgery
  Measure the rate of R0 resection with all margins microscopically clear.
Events Free Survival, EFS | Through study completion, an average of 1 year.
  Event-free survival was defined as the time from the date of randomization to the date of the first documented non-fatal event (worsening cardiac function, hospitalization for congestive heart failure, liver function impairment, liver cirrhosis, transformation to AML, as defined in the protocol), or death, whichever occurred first. Participants who did not experience a non-fatal event as of the time of data cut-off (end of study), as well as participants who did not experience a non-fatal event and stopped study participation before the data cut-off, were censored as specified in the protocol.
Overall Survival,OS | 5 years after inclusion
  Overall survival was the duration from the start of study treatment to death.
disease-free survival, DFS | 5 years after inclusion
  DFS is defined as the time interval between the date of random assignment and the date of the first documented evidence of relapse at any site or death related to cancer (including toxicity), whichever occurred first.
Disease Control Rate, DCR | 3 years after inclusion
  he Disease Control Rate (DCR) will be defined as the proportion of patients with a best overall response of CR, PR or Stable Disease (SD) (RECIST V1.1) 2 months after randomization
Objective Response Rate, ORR | 3 years after inclusion
  The Objective Response Rate (ORR) will be defined as the proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR) (RECIST V1.1)
Circulating tumor DNA, ctDNA | Before neoadjuvant therapy, before surgery, 1, 6, 12, 18, 24 months after surgery
  Blood will be drawn and tested for ctDNA

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] He W, Bai H, Lv J, Tang P, Hu T, Zhou H, Xiao W, Peng L, Liu G, Wang K, Fang Q, Qi Y, Liang L, Zheng X, Qing H, Chen Y, Zhou Y, Xie W, Han Y, Leng X. Neoadjuvant chemotherapy or chemoradiotherapy plus sintilimab versus neoadjuvant chemoradiotherapy for locally advanced oesophageal squamous cell carcinoma: a study protocol of a multicentre, randomised, controlled, phase III trial (SCIENCE study). BMJ Open. 2025 Jun 4;15(6):e095828. doi: 10.1136/bmjopen-2024-095828. PMID 40467307